09-07-2022

Clinical study protocol

Protocol title: "Randomized controlled trial comparing endoscopic balloon dila-

tion versus endoscopic stricturotomy for short strictures (< 3 cm) related to

**Crohn's disease (the BEST-CD trial)** 

**Primary Investigator.**"

Dr. PARTHA PAL

Asian Institute of Gastroenterology

6-3-331, Somajiguda, Hyderabad, 5000082

**Study description** 

**Brief Summary** 

Crohn's disease (CD) related strictures can be treated endoscopically by endoscopic

balloon dilation (EBD) or endoscopic stricturotomy (EST). EBD is is the established

endoscopic treatment for short strictures in Crohn's disease. However, roughly half

had recurrent symptoms and two third require surgery after EBD. ES have been used

initially for endoscopic treatment of patients for whom EBD was unsuccessful. Sub-

sequently it was shown that ES is a better modality for treating CD related strictures

(specially short and anastomotic strictures) than EBD lowering the risk of future

surgery and procedure related perforation albeit with an increased risk of bleeding. ES

was shown to be non-inferior to re-do surgery in chronic pouch anastomotic sinus in

ulcerative colitis (UC) and ileocolic anastomotic strictures in CD thus reducing surgi-

cal morbidity. However, these two modalities have not been compared in a random-

ized controlled manner. We aimed to compare the two endoscopic treatments with re-

gard to clinical success, need for surgery or additional endoscopic procedure and safe-

09-07-2022

ty in patients with CD who have short (<3 cm), predominantly fibrotic stenosis excluding those in the small bowel not accessible by endoscope/colonoscopy.

| <b>Condition or disease</b> | Intervention or treatment |
|-----------------------------|-------------------------------------------|
| Crohn's disease | Intervention: Endoscopic balloon dilation |
| | Intervention: Endoscopic stricturotomy |

# **Detailed description**

**Study design:** Single centre, open-label, randomized trial to be done in Asian Institute of Gastroenterology, India

**Study population:** All eligible consecutive patients with CD who developed DEnova or anastomotic strictures will be included.

### **Study settings:**

The proposed study would be conducted in a high volume tertiary GI centre (Asian Institute of Gastroenterology) performing nearly more than 200 EBD/ES procedures per year with an well established inflammatory bowel disease (IBD) registry with more than 7000 IBD patients under follow up.

The study will be conducted after approval by the institutional ethics committee. Written informed consent would be taken from each participants and the study would conform to the 1975 Declaration of Helsinki ethical guidelines.

**Data collection:** A survey administration software (google forms) would be used to collect the participant data (age, sex, ethnicity, clinical features, smoking status, details of CD diagnosis, disease phenotype, extra intestinal manifestations, family history, history of intestinal resection, details of stricture diagnosis, details of stricture: degree, number, location, radiological finding: concurrent abscess, fistula, enhancement;

09-07-2022

drug history for CD, procedural details: technical success, symptomatic improvement, endoscopic improvement, stricture related emergency visit or hospitalization, complications, subsequent need for additional endoscopic procedures or surgery upto a follow up of 1 year). Follow-up details would be collected via physical visit or telephonic communication.

Technique and instruments: EBD procedures will be performed with wire guided CRE pneumatic balloon (controlled radial expansion balloon, Boston scientific, Marlborough, MA, USA 0of various sizes based on tightness of the stricture (10-12 mm, 12-15 mm, 15-18 mm, 18-20 mm) with graded dilation with inflation pressures varying from 3-8 ATM pressure. Balloon was inflated for at least 2 minutes and slowly deflated. For mild ooze post EBD, balloon tamponade will also done with the same balloon. A maximum of two sessions of dilation will be allowed with a minimum interval of 15-30 days between them. Additional EBD sessions would be considered as additional endoscopic procedure for the purpose of the study.

Endoscopic stricturotomy would be done using a needle knife/insulted tip (IT) knife with the following electrocautery settings: Endocut Q (effect 3, cut duration 1, cut interval 3) as per by global IIBD group consensus.

**Definitions:** Technical success for EBD was defined as ability to perform the EBD procedure. Scope passage after EBD/stricturotomy was assessed as a separate outcome which was defined as passage of endoscope through the area where EBD/ES was performed. This included colonoscopy for colonic/pouch strictures, endoscope for upper GI and duodenal strictures and an endoscope: motorized spiral or single balloon enteroscopy for small bowel strictures except those in terminal ileum. Clinical

Study No: IBD-001

09-07-2022

Version No: 01 Date:

success in EBD/ES was defined as clinical improvement in symptoms (pain/ intesti-

nal, gastric outlet or colonic obstruction symptoms) after the procedure. Sustained

clinical success was defined as absence of obstructive symptoms at 1 year follow up.

Major adverse events were defined as perforation, bleeding requiring transfusion or

any procedure related prolongation of hospitalization period or an endoscopic, radio

logic or surgical intervention. Minor adverse events were bleeding not requiring blood

transfusion, post procedural pain and any other self limiting complication (e.g., sore

throat after spiral enteroscopy) which does not warrant prolongation of hospital stay.

Adverse events will be recorded for all the patients; events were considered associat-

ed to be with the procedure when a causal association was possible, probable, or defi-

nite. Recurrence of symptoms would be defined as re-emergence of symptoms for

which the procedure was initially performed.

Sample size

Based on previous retrospective study, symptomatic improvement with EST and EBD

(9.5% and 33.5% respectively, the estimated sample size is total 90 (45 in each group)

keeping type 1 error as 0.05 and power as 80%.

Randomization

Patients will be randomly assigned (1:1) to receive either EBD (EBD group) or EST

(EST group) using a digital en-block randomization system (block size of four).

Data analysis

Statistical analysis: Statistical analysis would be done by using statistical package for

social sciences (SPSS, IBM, NY, USA). Chi-square/Fisher's exact test was used to

09-07-2022

compare categorical variables and Mann-Whitney test would used to compare contin-

uous variables between the two groups.P-value < 0.05 would be considered statistical-

ly significant

Timeline: 2 years

Recruitment of 100 CD patients with stenosis requiring EBD or EST over 1 years:

follow up over 1 year.

**Patient privacy** 

An organized database for the purpose of this study will be formed based on google

form with anonymize data set (i.e. name, address, and full post code will be removed,

together with any other information which, in conjunction with other data held by or

disclosed to the recipient, could identify the patient) which would be entered by clini-

cal research assistant.

Study design

**Study type:** Interventional (clinical trial)

**Estimated enrolment:** 100 patients

**Allocation:** Randomized

**Intervention model:** Parallel assignment

**Masking:** none (open label)

**Primary purpose:** Therapeutic

Official title: Randomized controlled trial comparing endoscopic balloon dilation

versus endoscopic stricturotomy for short strictures (< 3 cm) related to Crohn's dis-

ease (the BEST-CD trial)

**Estimated start date :** August - September 2022 (after ethical approval)

09-07-2022

**Estimated recruitment completion:** July - August 2023

**Estimated study completion date:** July - August 2023

# **Arms and interventions:**

| Arm | Intervention/treatment |
|---|---|
| Active comparator: | Intervention: Endoscopic balloon dilation |
| Confirmed Crohn's disease | EBD procedures will be performed with wire |
| with gastro-duodenal or ileo- | guided CRE pneumatic balloon (controlled radial |
| colonic short (<3 cm) | expansion balloon, Boston scientific, Marlborough, |
| strictures (both de novo and | MA, USA 0of various sizes based on tightness of |
| anastomotic) without prior | the stricture (10-12 mm, 12-15 mm, 15-18 mm, |
| history of endoscopic | 18-20 mm) with graded dilations with inflation |
| stricture therapy | pressures varying from 3-8 ATM pressure. Balloon |
| | was inflated for at least 2 minutes and slowly |
| | deflated. A maximum of two sessions of dilation |
| | will be allowed with a minimum interval of 15-30 |
| | days between them. |

09-07-2022

**Intervention:** Endoscopic stricturotomy with or **Active comparator** Confirmed Crohn's disease without stricturoplasty with gastro-duodenal or ileo-Endoscopic stricturotomy would be done using colonic short (<3 cm) either a tri- ple-lumen needle-knife (Boston strictures (both de novo and Scientific, Marlborough, MA) or with a anastomotic) without prior electrosurgical IT knife2 (Olympus Medical history of endoscopic Systems, Tokyo, Japan) in the setting of ERCP stricture therapy Endocut on ERBE (USA Incorporated Surgical Systems, Marietta, GA) with the following electrocautery settings: Endocut Q (effect 3, cut duration 1, cut interval 3). Strictures will be incised in a circumferential or radial fashion until an adequate passage of the scope. Endoclips may be applied post stricturotomy to act as keep treated stricture open and to prevent delayed bleeding (referred as stricturoplasty). Choice of endoclips and decision to perform stricturoplasty would be at the discretion of endoscopist.

#### **Outcome measures**

### **Primary outcome measures**

To compare sustained clinical improvement post EBD and ES (%) (time frame :

09-07-2022

lyear): percentage of patients having no obstructive symptoms due to CD related

stenosis for which EBD/ES was performed for a period of 1 year

**Secondary outcome measures** 

1. To compare need for additional intervention (EBD/EST/Surgery) between EST and

EBD arm (%): the percentage of patients who require additional interventions for

CD related stenosis over period of 1 year

2. To compare technical success between EBD and ES (%): Percentage of patients in

whom endoscope is passable after EBD/ES

2. To compare stricture related visit to the emergency department after EST versus

EBD: percentage of patients visiting the emergency department for CD stenosis relat-

ed symptoms post EBD/ES over period of 1 year

3. To compare structure related hospitalization with EST versus EBD: percentage of

patients visiting undergoing hospitalization for CD stenosis related symptoms post

EBD/ES over period of 1 year

4. To compare complications related to EST versus EBD: Major adverse events will

be defined as perforation, bleeding requiring transfusion or any procedure related pro-

longation of hospitalization period or an endoscopic, radio logic or surgical interven-

tion. Minor adverse events were bleeding not requiring blood transfusion, post pro-

cedural pain and any other self limiting complication which does not warrant prolon-

gation of hospital stay. Adverse events were considered associated to be with the pro-

cedure when a causal association was possible, probable, or definite.

Eligibility criteria

Ages eligible for the study: 18 Years to 65 Years (Adult, Older Adult)

Sexes eligible for the study: all

Study No: IBD-001 09-07-2022 Version No: 01 Date:

Accepts healthy volunteer: no

| Authors | Patients<br>(N) | Location | Technical<br>Success | Adverse events |
|---|---|---|---|---|
| Lan et al 2015 | 85 | Multiple locations | 100% | 3.7% |
| Lan et al 2018 | 21 | Anastomotic | 100% | 8.8% |
| Lan et al 2019 | 35 | Anastomotic | 100% | 10.2% |
| Zhang et al 2019 | 49 | Multiple locations | 100% | 4.7% |
| Lan et al 2019 | 40 | Pouch Inlet | 100% | 4.7% |
| Kochhar G 2020 | 11 | Multiple locations | 92% | 9.0% |
| Lan et al 2020 | 13 | Terminal ileum | 100% | 6.9% |
| Moroi et al 2020 | 5 | Anastomotic | 100% | 20% |

# Criteria

| Outcome | | Stricturotomy<br>(n=21) | Balloon Dilation<br>(n=154) | P value |
|---|---|---|---|---|
| Follow-up time, year | | 0.8 (0.1–1.6) | 4.0 (0.8-6.9) | < 0.001 |
| Age at procedure, year | | 43.3 ± 14.5 | 42.8 ± 13.4 | 0.76 |
| Duration from last surgery to procedure, year | | 6.4 (1.7-16.4) | 7.8 (3.6-13.3) | 0.56 |
| Duration from CD diagnosis to procedure, year | | 19.6 (11.4-8.1) | 16.6 (9.9-25.8) | 0.85 |
| Immediate technical success | | 21 (100.0%) | 147 (89.5%) | 0.25 |
| Symptomatic improvement | | 8/11 (72.7%) | 59/103(45.4%) | 0.08 |
| Endoscopic improvement | | 8/17 (47.1%) | 57/163(35.0%) | 0.32 |
| Escalation of drug after procedure | | 13 (61.9%) | 53 (32.3%) | 0.09 |
| Additional endoscopic therapy (EBD or ES) | | 6 (28.6%) | 98 (59.8%) | 0.85 |
| Outcome | | Stricturetomy<br>(N=21) | Balloon Dilation<br>(n=164) | P value |
| Outcome Disease related emergency depart | artment visits | | | P value<br>0.74 |
| | artment visits<br>Per Patients | (N=21) | (n=164) | |
| Disease related emergency depart | | (N=21)<br>2 (9.5%) | (n=164)<br>40 (24.4%) | 0.74 |
| Disease related emergency depart | Per Fatients | (N=21)<br>2 (9.5%)<br>1 (2.0) | (n=164)<br>40 (24.4%)<br>34 (20.7%) | 0.74 |
| Disease related emergency depa<br>Stricture-related | Per Fatients | (N=21)<br>2 (9.5%)<br>1 (2.0)<br>4/11 (36.4%) | (n=164)<br>40 (24.4%)<br>34 (20.7%)<br>78/104(75.0%) | 0.74<br>0.33<br>0.001 |
| Disease related emergency depa<br>Stricture-related | Per Fatients<br>Per visit | (N=21)<br>2 (9.5%)<br>1 (2.0)<br>4/11 (36.4%)<br>7 (33.3%) | (n=164)<br>40 (24.4%)<br>34 (20.7%)<br>78/104(75.0%)<br>40 (24.4%) | 0.74<br>0.33<br>0.001<br>0.93 |
| Disease related emergency depa<br>Stricture-related | Per Patients Per visit Per Patients | (N=21)<br>2 (9.5%)<br>1 (2.0)<br>4/11 (36.4%)<br>7 (33.3%)<br>1 (4.8%) | (n=164) 40 (24.4%) 34 (20.7%) 78/104(750%) 40 (24.4%) 33 (20.1%) | 0.74<br>0.33<br>0.001<br>0.93<br>0.16 |
| Disease related emergency departments of the Stricture-related Disease related hospitalization Stricture related | Per Patients Per visit Per Patients | (N=21)<br>2 (9.5%)<br>1 (2.0)<br>4/11 (36.4%)<br>7 (33.3%)<br>1 (4.8%) | (n=164) 40 (24.4%) 34 (20.7%) 78/104(750%) 40 (24.4%) 33 (20.1%) | 0.74<br>0.33<br>0.001<br>0.93<br>0.16 |
| Disease related emergency depa<br>Stricture-related Disease related hospitalization Stricture related Complication | Per Patients Per Patients Per visit | (N=21)<br>2 (9.5%)<br>1 (2.0)<br>4/11 (36.4%)<br>7 (33.3%)<br>1 (4.8%)<br>2/12 (16.7%) | (n=164) 40 (24.4%) 34 (20.7%) 78/104(75.0%) 40 (24.4%) 33 (20.1%) 57/102(55.9%) | 0.74<br>0.33<br>0.001<br>0.93<br>0.16<br>0.35 |
| Disease related emergency depa<br>Stricture-related Disease related hospitalization Stricture related Complication | Per Patients Per Patients Per visit Per patients | (N=21)<br>2 (9.5%)<br>1 (2.0)<br>4/11 (36.4%)<br>7 (33.3%)<br>1 (4.8%)<br>2/12 (16.7%) | (n=164) 40 (24.4%) 34 (20.7%) 78/104(75.0%) 40 (24.4%) 33 (20.1%) 57/102(55.9%) | 0.74<br>0.33<br>0.001<br>0.93<br>0.16<br>0.35 |
| Disease related emergency departments of the Stricture-related Disease related hospitalization Stricture related Complication Perforation | Per Patients Per Patients Per visit Per patients Per patients Per procedures | (N=21) 2 (9.5%) 1 (2.0) 4/11 (36.4%) 7 (33.3%) 1 (4.8%) 2/12 (16.7%) 0/21 (0.0%) 0/45 (0.0%) | (n=164) 40 (24.4%) 34 (20.7%) 78/104(750%) 40 (24.4%) 33 (20.1%) 57/102(55.9%) 4/164 (2.4%) 5/478 (1.1%) | 0.74<br>0.33<br>0.001<br>0.93<br>0.16<br>0.35 |

Version No: 01

Study No: IBD-001 09-07-2022 Date:



5-year surgery-free survival curve after treated with endoscopic stricturotomy (ES) versus endoscopic balloon dilation (EBD).





### **Inclusion Criteria:**

Primary confirmed diagnosis of CD with obstructive symptoms

1) Gastro-duodenal and ileo-colonic strictures (both de novo and anastomotic strictures)

09-07-2022

2) Short strictures (<3 cm)

- 3) Fibrotic or mixed stricture (predominantly fibrotic)
- 4) Strictures treated with either EST or EBD.

#### **Exclusion Criteria:**

- 1. No established diagnosis of CD;
- 2. No endoscopic therapy; and
- 3. A combination therapy of EST and EBD at the onset
- 4. Small bowel CD related stricture requiring enteroscopy guided dilation
- 5. Predominantly ulcerated strictures (mixed or pure ulcerated strictures)
- 6. Long strictures (>3 cm)
- 7. Pediatric Patients (<18 years)
- 8. Pregnant or lactating mother
- 7. Not willing to participate

Studies on ESTST vs EBD CD related anastomotic strictures

# **Experience of the key project personnel**

Dr. PARTHA PAL, MD, DNB, MRCP (UK)): Consultant Gastroenterologist with special interest in IBD research at IBD Center, Asian Institute of Gastroenterology,

09-07-2022

Hyderabad India. He runs the IBD Clinic at the AIG, Somajiguda unit with an established IBD registry and is actively involved in research in the field of IBD with numerous publications. He is also a co-investigator of numerous clinical trials in IBD.

## **Declaration of Investigator**

I have read and understood all sections of the protocol entitled "Randomized controlled trial comparing endoscopic balloon dilation versus endoscopic stricturotomy for short strictures (< 3 cm) related to Crohn's disease (the BEST-CD trial)" in the accompanying investigator's brochure. I agree to supervise all aspects of the protocol and to conduct the clinical investigation in accordance with the Final Protocol Version including country specific dated—the International Council for Harmonization harmonized tripartite guideline E6(R2): Good Clinical Practice and the Declaration of Helsinki (WMA2013), and all applicable government regulations. I will not make changes to the protocol before consulting implement protocol changes without independent ethics committee approval except to eliminate an immediate risk to patients. I agree to perform the procedure only to patients under my personal supervision or the supervision of a sub-investigator. Confidentiality will be protected. Patient identity will not be disclosed to third parties or appear in any study reports or publications.

| Signature of Principal Investigator | Date |
|----------------------------------------|------|
| Printed Name of Principal Investigator | |